CLINICAL TRIAL: NCT01324063
Title: A Randomized Phase III Study of Intensive Consolidation With High Dose Cytosine Arabinoside in Acute Myelogenous Leukemia (AML-8B)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-06864; EORTC-06864
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia | interventions — sargramostim; Amsacrine; Cytarabine; Daunorubicin

INTERVENTIONS:
Biological: sargramostim
Drug: amsacrine
Drug: cytarabine
Drug: daunorubicin hydrochloride
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Patient abstract not available

PURPOSE: Patient abstract not available

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the value (in terms of disease-free survival and overall survival) of short intensive consolidation with high-dose cytosine arabinoside in patients with acute myelogenous leukemia who achieve complete remission after induction with daunorubicin and cytosine arabinoside. II. Assess the toxicity and resulting quality of life associated with consolidation with high-dose cytosine arabinoside compared with conventional consolidation/maintenance treatment. III. Determine whether addition of granulocyte-macrophage colony stimulating factor (GM-CSF) to Induction chemotherapy can improve therapeutic results through activation of leukemic cells into the cell cycle and/or acceleration of hematopoietic recovery (objective added 08/90). IV. Determine indirectly whether autologous bone marrow therapy is better than conventional consolidation/maintenance or high-dose cytosine arabinoside by comparing results from protocol EORTC-06863 (AML 8 A).

OUTLINE: Patients with normal kidney function are randomized on Arms A-D for Induction (patients whose serum creatinine is more than 1.5 x the upper limit of normal are nonrandomly assigned to Arm A). Following Induction, patients achieving CR are randomized to Arms I and II. Induction: Arm A: 2-Drug Combination Chemotherapy. Daunorubicin, Daunomycin, DNM, DNR, NSC-82151; Cytosine arabinoside, ARA-C, NSC-63878. Arm B: 2-Drug Combination Chemotherapy plus Growth Factor Therapy. DNM; ARA-C; plus Granulocyte-Macrophage Colony Stimulating Factor (Sandoz), GM-CSF. GM-CSF on days 0 through 7. Arm C: 2-Drug Combination Chemotherapy with Hematologic Toxicity Attenuation. DNM; ARA-C; GM-CSF. GM-CSF from end of chemotherapy through day 28. Arm D: 2-Drug Combination Chemotherapy plus Growth Factor Therapy and Hematologic Toxicity Attenuation. DNM; ARA-C; GM-CSF. GM-CSF on days 0 through 28. Arm I: Intensive Consolidation: 2-Drug Combination Chemotherapy followed by 2-Drug Combination Chemotherapy. High-dose ARA-C, HDARA-C; Acridinylanisidide, m-AMSA, AMSA, NSC-249992; followed by HDARA-C; DNR. Arm II: Standard Consolidation/Maintenance: 2-Drug Combination Chemotherapy. ARA-C; DNR.

PROJECTED ACCRUAL: A minimum of 157 patients will be required; with an expected entry rate of 40 patients per year, patient entry is expected to take 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed, untreated acute myelogenous leukemia (AML), as follows: Any cytological type according to the FAB classification At least 30% blast cells in bone marrow smear required Secondary acute leukemia eligible, i.e.: AML cured Hodgkin's disease or other malignancy AML following exposure to alkylating agents or radiation The following are specifically excluded: Blast crisis of chronic myeloid leukemia Leukemia supervening after other myeloproliferative disease Leukemia supervening after overt myelodysplastic disorder (e.g., refractory anemia with excess blasts) of more than 6 months' duration

PATIENT CHARACTERISTICS: Age: 45-60 Patients 10-45 are eligible for EORTC-06863 Performance status: Not specified Hematopoietic: Not specified Hepatic: No severe concomitant hepatic disease Renal: No severe concomitant renal disease Cardiovascular: No severe concomitant cardiac disease Other: No severe concomitant neurological disease No other progressive malignant disease

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior therapy Chemotherapy: No prior chemotherapy Endocrine therapy: No more than 7 days of corticosteroids for AML Radiotherapy: No prior radiotherapy Surgery: Not applicable

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 1986-11; Primary Completion 1994-06 (Actual)

PRIMARY OUTCOMES:
Disease-free survival and overall survival in patients who achieve complete remission after induction
Toxicity
Quality of life
Improved therapeutic results as measured by activation of leukemic cells into the cell cycle and/or acceleration of hematopoietic recovery
Relative efficacy of autologous bone marrow therapy

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Zittoun, MD, Study Chair — Hotel Dieu de Paris

REFERENCES:
- [Result] Zittoun R, Suciu S, Mandelli F, de Witte T, Thaler J, Stryckmans P, Hayat M, Peetermans M, Cadiou M, Solbu G, Petti MC, Willemze R. Granulocyte-macrophage colony-stimulating factor associated with induction treatment of acute myelogenous leukemia: a randomized trial by the European Organization for Research and Treatment of Cancer Leukemia Cooperative Group. J Clin Oncol. 1996 Jul;14(7):2150-9. doi: 10.1200/JCO.1996.14.7.2150. PMID 8683249